CLINICAL TRIAL: NCT07336394
Title: Multimodality Imaging (Cardiovascular Magnetic Resonance Imaging, Echocardiography, and Nuclear Medicine Imaging) in the Screening, Diagnosis and Risk Stratification of Rare Cardiomyopathies - a Multicenter Study
Brief Title: Precision Diagnosis and Risk Stratification of Rare Cardiomyopathies Based on Novel Cardiac Magnetic Resonance Techniques
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Anzhen Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Minjie Lu, Director of Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR-RareCM
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Danon Disease; Fabry Disease; Cardiac Amyloidosis; Noonan Syndrome; Cardiac Sarcoidosis; Glycogen Storage Disease; Idiopathic Cardiomyopathy
Keywords: cardiovascular magnetic resonance imaging; early diagnosis; prognosis; rare cardiomyopathies; nuclear medicine imaging; echocardiography
MeSH Terms: conditions — Glycogen Storage Disease Type IIb; Fabry Disease; Amyloid Neuropathies, Familial; Noonan Syndrome; Glycogen Storage Disease; Cardiomyopathies; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — data of radiology imaging, clinical study and laboratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is this study about? This research is focused on improving the care for people with rare heart muscle diseases, known as rare cardiomyopathies. These are uncommon conditions where the heart muscle becomes stiff, thick, or enlarged, making it harder for the heart to pump blood. Because they are rare, they can be difficult to diagnose and manage.

The investigators are testing new, advanced ways of using a heart scan called a Cardiac Magnetic Resonance (CMR). Participants can think of a CMR as a very powerful camera that takes detailed pictures of their heart without using radiation.

What is the study trying to learn? Better Diagnosis: The investigators want to see if these new scanning techniques can help us identify these rare heart conditions more clearly and accurately. This means patients could get a correct diagnosis sooner.

Personalized Risk Assessment: The investigators want to see if the scan can help us understand the future risk for each patient better. For example, can it help predict which patients are more likely to have a heart rhythm problem or need specific treatments? This helps doctors create a care plan that is tailored just for participants.

What does this mean for participants? If participants choose to take part, they will undergo a CMR scan that uses these new techniques. By participating, they will be helping us find better ways to diagnose and care for people with their condition in the future. The goal is to turn uncertainty into clearer, more personalized information for patients and families.

DETAILED DESCRIPTION:
Study Objective:

This study aims to validate and apply novel Cardiac Magnetic Resonance (CMR) imaging biomarkers to improve the diagnostic precision and risk stratification of rare cardiomyopathies (e.g., cardiac amyloidosis, Fabry disease, Danon disease, Noonan disease).

Clinical Problem:

Rare cardiomyopathies are often challenging to diagnose due to overlapping phenotypic features with more common disorders and their heterogeneous presentation. Current risk stratification tools are imperfect, leading to delays in diagnosis and suboptimal timing of interventions.

Methodology & Innovation:

The study will employ advanced CMR techniques that move beyond standard volumetric and functional assessment. This includes, but is not limited to:

T1/T2 Mapping: For quantitative tissue characterization to detect diffuse fibrosis or edema without contrast.

Extracellular Volume (ECV) Fraction: To quantify the expansion of the extracellular space, a key marker in amyloidosis and other infiltrative diseases.

Feature Tracking Strain Analysis: To assess subtle myocardial deformation abnormalities that precede a decline in ejection fraction.

Late Gadolinium Enhancement (LGE) Pattern Refinement: For more precise characterization of scar and infiltration patterns.

Potential Impact for Clinical Practice:

Referral & Diagnosis: This research could provide more definitive, non-invasive diagnostic data, streamlining the referral pathway to specialist centers and reducing diagnostic odysseys for patients.

Risk Stratification: The novel biomarkers investigated have the potential to offer superior prognostic value compared to current clinical models. This can aid in identifying high-risk patients earlier, guiding decisions regarding device therapy (ICD) initiation or referral for advanced therapies.

Management: By providing a more detailed "tissue phenotype," the findings could help monitor disease progression and response to emerging targeted therapies more sensitively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a cardiac magnetic resonance examination since 2010 and have a suspicion of rare cardiomyopathy.

Exclusion Criteria:

* Severe arrhythmia;
* Severe primary cardiac valvular disease;
* Refuse to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received a cardiac magnetic resonance examination since 2010 and have a suspicion of rare cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of All-cause Death | 2-15 years
  the incidence of all-cause death
Incidence Rate of Cardiovascular Death | 2-15 years
  the incidence of cadridovascular death
Incidence Rate of Heart Transplantation | 2-15 years

SECONDARY OUTCOMES:
Incidence Rate of Hospitalization Due to Heart Failure | 2-15 years
Incidence Rate of Implantable cardioverter-defibrillator Implantation | 2-15 years
Incidence Rate of Pacemaker Implantation | 2-15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Our study data is applicable to other researchers with permmsion.

REFERENCES:
- [Result] Zhang Q, Li J, Lu M. Rare imaging phenotype of late gadolinium enhancement in a patient with anoctamin 5 mutation. Eur Heart J Case Rep. 2024 Nov 23;8(12):ytae626. doi: 10.1093/ehjcr/ytae626. eCollection 2024 Dec. No abstract available. PMID 39659467
- [Result] Yue X, Yang K, Lu M. A tale of two phenotypes: transition from hypertrophic to dilated cardiomyopathy in Danon disease. Eur Heart J Case Rep. 2024 Aug 26;8(9):ytae445. doi: 10.1093/ehjcr/ytae445. eCollection 2024 Sep. No abstract available. PMID 39290522
- [Result] Lv Y, Li JH, Lu M. Glycogen storage disease type IIIa: a rare cause of myocardial hypertrophy with multisystem involvement. Eur Heart J Cardiovasc Imaging. 2025 Mar 27;26(4):764. doi: 10.1093/ehjci/jeae328. No abstract available. PMID 39700428
- [Result] He J, Xu J, Chen L, Ji K, Fan X, Zhao S, Lu M. Clinical features and cardiovascular magnetic resonance characteristics in Danon disease. Clin Radiol. 2020 Sep;75(9):712.e1-712.e11. doi: 10.1016/j.crad.2020.04.012. Epub 2020 Jun 1. PMID 32499120
- [Result] Gu X, Dai L, Lu M. Mucolipidosis III: a rare phenocopy of inherited metabolic cardiomyopathy. Eur Heart J. 2024 Nov 8;45(42):4548. doi: 10.1093/eurheartj/ehae636. No abstract available. PMID 39344930